CLINICAL TRIAL: NCT02327546
Title: An Open-Label, Randomized, Single-Dose Study to Evaluate the Effects of 325 mg Ferrous Sulfate Tablet (65 mg Iron) on the Pharmacokinetics of 450 mg Dose of AKB-6548 in Healthy Male Volunteers.
Brief Title: Effects of Ferrous Sulfate on the Pharmacokinetics of AKB-6548
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AKB-6548-CI-0012
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Anemia; Chronic kidney disease; CKD; Chronic renal insufficiency; Renal impairment; Ferrous sulfate; Iron; Drug-drug interaction; End stage renal disease; Dialysis; Erythropoietin; Oral anemia treatment; Hypoxia-induciable factor; HIF; Hypoxia-induciable factor prolyl-hydroxylase inhibitor; HIF-PHI
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Renal Insufficiency; Kidney Failure, Chronic | interventions — vadadustat; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AKB-6548 (Experimental): AKB-6548
  Interventions: Drug: AKB-6548
- AKB-6548 plus Ferrous Sulfate (Experimental): AKB-6548 plus ferrous sulfate
  Interventions: Drug: AKB-6548; Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: AKB-6548
Drug: Ferrous Sulfate
  Arms: AKB-6548 plus Ferrous Sulfate

SUMMARY:
The primary purpose of this study is to assess the single-dose bioavailability of AKB-6548 with ferrous sulfate relative to AKB-6548 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects 18 to 55 years of age with a body mass index between 18 and 30 kg/m2
* Participants and their partners must use a highly effective form of contraception during the study and for 1 month following discharge from the Clinical Research Unit (CRU)
* Subjects must discontinue all iron preparations for 14 days prior to study drug administration

Exclusion Criteria:

* Current or past history of cardiovascular, cerebrovascular, pulmonary, renal or liver disease
* Positive serology results for HBsAg, HCV, and HIV at Screening
* Renal impairment (estimated glomerular filtration rate (eGFR) of <65mL/min)
* Known active cancer (except non-melanoma skin cancer) or history of chemotherapy use within the previous 24 months
* Current or past history of gastric or duodenal ulcers or other diseases of the GI tract (including gastric bypass surgeries) that could interfere with absorption of study drug
* Subjects with a known history of smoking and/or have used nicotine or nicotine-containing products within the past 6 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
PK parameters of AKB-6548: Maximum plasma concentration (Cmax) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548: Area under the curve from time 0 until the last quantifiable concentration (AUC [last]) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548: Area under the concentration-time curve from 0 to infinity (AUCinf) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose

SECONDARY OUTCOMES:
PK parameters of AKB-6548: Time to maximum plasma concentration (Tmax) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548: Terminal elimination rate constant (λz) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548: Plasma half life (t1/2) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548: Apparent total systemic clearance (CL/F) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548: Apparent volume of distribution during the terminal elimination phase (VzF) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548 metabolites: Maximum plasma concentration (Cmax) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548 metabolites: Time to maximum plasma concentration (Tmax) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548 metabolites: Terminal elimination rate constant (λz) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548 metabolites: Plasma half life (t1/2) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548 metabolites: Area under the curve from time 0 until the last quantifiable concentration (AUC [last]) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
PK parameters of AKB-6548 metabolites: Area under the concentration-time curve from 0 to infinity (AUCinf) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
Ratio of metabolite to parent drug for maximum plasma concentration (Cmax) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
Ratio of metabolite to parent drug for are under the curve from time 0 until the last quantifiable concentration (AUC [last]) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose
Ratio of metabolite to parent drug for area under the concentration-time curve (AUC) | Multiple timepoint evaluations from pre-dose to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (1):
- Kalamazoo, Michigan, United States